CLINICAL TRIAL: NCT00826111
Title: The Effects of Eszopiclone and Lexapro on Prefrontal Glutamate and GABA in Depression With Co-morbid Anxiety and Insomnia: A Proton MRS Study
Brief Title: The Effects of Eszopiclone and Lexapro on Prefrontal Glutamate and GABA in Depression With Anxiety and Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00427
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Results first posted 2012-06-29 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Depression; Anxiety; Insomnia
Keywords: Magnetic Resonance Spectroscopy; Glutamate; Glutamine; GABA; Lexapro; Lunesta; Escitalopram; Eszopiclone
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eszopiclone (Active Comparator): Lexapro for 10 weeks together with eszopiclone.
  Interventions: Drug: Eszopiclone
- Placebo (Placebo Comparator): Lexapro for 10 weeks together with placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone — Subjects receive 10 mg escitalopram daily for four weeks and 10 or 20 mg for an additional six weeks. Subjects also receive 3 mg eszopiclone.
  Other Names: Lunesta
  Arms: Eszopiclone
Drug: Placebo — Subjects receive 10 mg of escitalopram daily for four weeks followed by 10 or 20 mg for an additional six weeks. Subjects also receive placebo for eszopiclone.
  Arms: Placebo

SUMMARY:
The study examined the effects of adding the sleep aid eszopiclone to Lexapro on mood and levels of the neurotransmitters glutamate, glutamine, and GABA in women with depression, anxiety, and insomnia. Specifically, the objective was to determine the role of glutamate, glutamine, and GABA in mediating the response the to the combined treatment. The hypothesis was that levels of glutamine and glutamate will be increased in women receiving eszopiclone compared to those receiving placebo. The antidepressant effect of the medication combination and its effect on sleep status was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 to 55 years and regularly menstruating.
* Meets DSM-IV criteria for unipolar major depression.
* Insomnia severity index score > 10.
* Hamilton Anxiety scale score > 15.
* Hamilton Depression scale score > 17.
* Capable of providing informed consent.
* Has an established residence and phone.

Exclusion Criteria:

* Meets DSM-IV criteria for schizophrenia, schizoaffective disorder or other axis I or II diagnosis except co-morbid anxiety disorder and insomnia.
* Actively abusing substances or alcohol; or has met DSM-IV criteria for substance dependence in the past month.
* Pregnancy.
* Use of benzodiazepines or other sedative-hypnotics, beta blockers, calcium channel blockers, antidepressants, antipsychotic medications, lithium or other medication which in the opinion of the investigator could alter glutamate or GABA activity in the brain.
* A medical condition, which in the opinion of the investigator could possibly affect the individual's brain levels of Glu and GABA.
* Participation in a research protocol that included administration of medication within the past 3 months.
* Cigarette smoking.
* Subject has known allergic sensitivity to any of the study to escitalopram, eszopiclone or zopiclone.
* Clinically significant suicidal ideation or risk of suicide as evidenced by formulation of a plan or steps taken to act on those feelings.
* History of clinically significant hepatic impairment.
* Subject is taking a potent cytochrome p450 3A4 inhibitor medication (ritonavir, nelfinavir, indinavir, erythromycin, clarithromycin, troleandomycin, ketoconazole, itraconazole) and is unwilling or it is clinically contraindicated to stop the medication.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2007-08; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Henry, MD, Principal Investigator — Steward St. Elizabeth's Medical Center of Boston, Inc.
Locations (1):
- Steward St. Elizabeth's Medical Center of Boston, Inc., Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from September 2008 until October 2010. Participants were recruited by advertising in the community.
Pre-assignment Details: Enrolled participants were excluded before assignment to groups if they had another co-morbid psychiatric diagnosis, a medical condition that could affect glutamate or GABA levels, a clinical presentation that was not consistent with a diagnosis of major depressive disorder, or rating scale scores below the minimum for inclusion.
Groups:
- Placebo: Escitalopram with placebo
Period: Overall Study
Arm/Group | Eszopiclone | Placebo
Started | 14 | 5
Completed | 7 | 3
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eszopiclone | Placebo | Total
Number analyzed (Participants) | 14 | 5 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 5 | 19
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.8 (7.5) | 25.4 (5.0) | 28.6 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Anterior Cingulate Cortex Glutamine From Baseline to Week 1.
Description: Glutamine levels were measured by single voxel magnetic resonance spectroscopy. In order to normalize the data, the glutamine values were expressed as a ratio to levels of creatine, since creatine levels are not expected to vary significantly.
Time Frame: baseline and 1 week
Population: Participants who had usable MRS data from both the baseline and week 1 scans were included in the analysis. Participants whose data was considered unreliable were excluded.
Measure: Mean (Standard Deviation); unit: ratio (glutamine to creatine)
Groups:
- Eszopiclone: Open label escitalopram for 10 weeks together with 3 mg eszopiclone for eight weeks followed by placebo for two weeks.
- Placebo: Open label escitalopram for 10 weeks together with placebo for 10 weeks.
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 10 | 4
ratio (glutamine to creatine) | 0.00059 (0.096) | 0.00908 (0.088)
Statistical Analysis 1: Comparison: Eszopiclone vs Placebo; Test type: Superiority or Other; p = 0.88, t-test, 2 sided; Mean Difference (Final Values) = 0.0085, 95% CI 2-sided [-0.1390 to .01220], Standard Error of Mean .0534

2. Primary Outcome: Change in Thalamic Glutamine From Baseline to Week 1
Description: Glutamine levels were measured by single voxel magnetic resonance spectroscopy in the left thalamus. In order to normalize the data, the glutamine values were expressed as a ratio to levels of creatine, since creatine levels are not expected to vary significantly.
Time Frame: baseline and 1 week
Population: Participants were included in the analysis if they had usable spectroscopy data from baseline and week 1 and were not considered to have any confounding issues such as an abnormal structural MRI.
Measure: Mean (Standard Deviation); unit: ratio (glutamine to creatine)
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 8 | 3
ratio (glutamine to creatine) | -0.6639 (0.292) | -0.3551 (0.076)
Statistical Analysis 1: Comparison: Eszopiclone vs Placebo; Test type: Superiority or Other; p = 0.79, t-test, 2 sided; Mean Difference (Final Values) = -0.031, 95% CI 2-sided [-0.286 to 0.224], Standard Error of Mean 0.112

3. Secondary Outcome: Change in Anterior Cingulate Cortex Glutamate From Baseline to Week 1
Description: Glutamate levels were measured in the anterior cingulate cortex using single voxel magnetic resonance spectroscopy. In order to normalize the data, the glutamate values were expressed as a ratio to levels of creatine, since creatine levels are not expected to vary significantly.
Time Frame: baseline and 1 week
Measure: Mean (Standard Deviation); unit: ratio (glutamate to creatine)
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 10 | 4
ratio (glutamate to creatine) | -0.0066 (.0148) | 0.215 (.0239)
Statistical Analysis 1: Comparison: Eszopiclone vs Placebo; Test type: Superiority or Other; p = 0.16, t-test, 2 sided; Mean Difference (Final Values) = -.0222, 95% CI 2-sided [-0.580 to .0136], Standard Error of Mean .0128

4. Secondary Outcome: Change in Thalamic Glutamate From Baseline to Week 1
Description: Glutamate levels were measured in the left thalamus using single voxel magnetic resonance spectroscopy. In order to normalize the data, the glutamate values were expressed as a ratio to levels of creatine, since creatine levels are not expected to vary significantly.
Time Frame: baseline and 1 week
Measure: Mean (Standard Deviation); unit: ratio (glutamate to creatine)
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 8 | 3
ratio (glutamate to creatine) | -0.0016 (0.287) | -0.7715 (0.874)
Statistical Analysis 1: Comparison: Eszopiclone vs Placebo; Test type: Superiority or Other; p = 0.29, t-test, 2 sided; Mean Difference (Final Values) = 0.710, 95% CI 2-sided [-1.35 to 2.77], Standard Error of Mean 0.515

5. Secondary Outcome: Change in Anterior Cingulate Cortex GABA From Baseline to Week 1
Description: GABA levels were measured in the anterior cingulate cortex using single voxel magnetic resonance spectroscopy. In order to normalize the data, the GABA values were expressed as a ratio to levels of creatine, since creatine levels are not expected to vary significantly.
Time Frame: baseline and 1 week
Measure: Mean (Standard Deviation); unit: ratio (GABA to creatine)
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 10 | 4
ratio (GABA to creatine) | 0.0013 (0.008) | -0.0036 (0.008)
Statistical Analysis 1: Comparison: Eszopiclone vs Placebo; Test type: Superiority or Other; p = 0.37, t-test, 2 sided; Mean Difference (Final Values) = 0.0048, 95% CI 2-sided [-0.0077 to 0.0174], Standard Error of Mean 0.005

6. Secondary Outcome: Change in Thalamic GABA From Baseline to Week 1
Description: GABA levels were measured in the left thalamus using single voxel magnetic resonance spectroscopy. In order to normalize the data, the GABA values were expressed as a ratio to levels of creatine, since creatine levels are not expected to vary significantly.
Time Frame: baseline and 1 week
Measure: Mean (Standard Deviation); unit: ratio (GABA to creatine)
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 9 | 4
ratio (GABA to creatine) | -0.0002 (0.0115) | -0.0058 (0.0033)
Statistical Analysis 1: Comparison: Eszopiclone vs Placebo; Test type: Superiority or Other; p = 0.21, t-test, 2 sided; Mean Difference (Final Values) = 0.0056, 95% CI 2-sided [-0.0037 to 0.1481], Standard Error of Mean 0.0042

7. Secondary Outcome: Change in Hamilton Depression Rating Scale Score From Baseline to Week 10
Description: The Hamilton Depression Rating Scale is a 21 item scale that assesses symptoms of depression with items rated on a scale of 0-4 or 0-2. The total score range is 0 to 65. A score of 7 or lower is generally considered to be an absence of depressive symptoms. A score of 18 was considered to be the cut-off for enrollment in this study, as this indicates clinically significant depression. A higher score represents greater severity of depressive symptoms.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 10 | 4
scores on a scale | -13.4 (8.26) | -20.75 (5.91)
Statistical Analysis 1: Comparison: Eszopiclone vs Placebo; Test type: Superiority or Other; p = 0.10, t-test, 2 sided; Mean Difference (Final Values) = 7.35, 95% CI 2-sided [-1.76 to 16.46], Standard Error of Mean 3.94

8. Secondary Outcome: Change in Hamilton Anxiety Rating Scale Score From Baseline to Week 10
Description: The Hamilton Anxiety Rating Scale is a 14 item ordinal scale that assesses symptoms of anxiety with ratings from 0-4. The score range is 0 to 56, with a higher score indicating higher levels of anxiety. A score of 15 was designated as the cut-off for enrollment in the study.
Time Frame: baseline and 10 weeks
Population: Participants who completed 10 weeks and one participant who completed 6 weeks (using last observation carried forward) were included in this analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Eszopiclone: Escitalopram for 10 weeks together with eszopiclone.
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 8 | 3
scores on a scale | -11.4 (7.31) | -12 (6.68)
Statistical Analysis 1: Comparison: Eszopiclone vs Placebo; Test type: Superiority or Other; p = 0.89, t-test, 2 sided; Mean Difference (Net) = 0.6, 95% CI 2-sided [-9.31 to 10.51], Standard Error of Mean 4.06

9. Secondary Outcome: Change in Insomnia Severity Index Score From Baseline to Week 10
Description: The Insomnia Severity Index is a 7 item scale that assesses difficulty sleeping and effect on quality of life with item scores from 0-4. The total score range is 0 to 28 with higher scores indicating higher levels of impairment and distress.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 10 | 4
scores on a scale | -11.2 (8.30) | -9.5 (5.45)
Statistical Analysis 1: Comparison: Eszopiclone vs Placebo; Test type: Superiority or Other; p = 0.66, t-test, 2 sided; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-10.31 to 6.91], Standard Error of Mean 3.78

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at all study visits which occurred every one to two weeks.
Arm/Group | Eszopiclone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/5
Other Adverse Events (participants affected / at risk) | 3/14 | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eszopiclone (N=14) | Placebo (N=5)
jaw pain (General disorders) | 1 (1) | 0 (0)
somnolescence (General disorders) | 2 (2) | 0 (0)
MRI abnormality (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Withdrawal of support by the funding sponsor due to other priorities resulted in a very small sample size with a small placebo group. Participant withdrawal and unusable data explains discrepancies in subject numbers in some analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No